CLINICAL TRIAL: NCT01624818
Title: Coping With Physical Activity and Psychosocial Challenges in Children With Heart Disease at Geilomo Childrens Hospital
Brief Title: Active With Heart Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 268289
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Heart Disease
Keywords: coping; physical activity; psychosocial; children; heart disease; habilitation
MeSH Terms: conditions — Heart Diseases; Motor Activity

ARMS (2):
- Group 2, 6-7 years (Experimental): 18 children (6-7 years) with heart disease participating in a rehabilitation programme in Geilomo childrens hospital
  Interventions: Behavioral: Cardiac habilitation program
- Group 1, 11-12 years (Experimental): 18 children(11-12 years) with heart disease participating in a rehabilitation programme at Geilomo childrens hospital.
  Interventions: Behavioral: Cardiac habilitation program

INTERVENTIONS:
Behavioral: Cardiac habilitation program — physical activity three weeks

SUMMARY:
Background: In Norway each year 130-150 children are born with heart disease that requires lifelong medical follow-up. Children with heart defects have reduced motor skills and reduced physical capacity compared with healthy peers. Increased knowledge in the children themselves and the general public, along with psychosocial interventions improve the child's ability to cope with the consequences of their disease. Descriptions of the experiences that Norwegian children with heart disease and their parents have about participation in rehabilitation programs is limited. Geilomo children's hospital has 75 years experience in rehabilitation of children with chronic illness, and started in 2005 to welcome children with heart disease. At present there is no rehabilitation institutions in Norway that has a special group programs for children with heart disease. Geilomo want to establish such a group for children aged 6-7 years and 11-12 years.

Main objective: The investigators will use of methods to learn more about the following:

Study 1: The purpose is to generate knowledge about how children with heart disease and their relatives experience participation in a rehabilitation program at Geilomo children's hospital.

Overarching question: How do children with heart disease and their guardians to participate in a rehabilitation program, and the impact of this on their daily life afterwards?

Study 2: The purpose is to help a) to give the children an increased level of activity in the home environment.

Question: Will children with heart disease increase their activity levels at home after a stay at Geilomo? 2b) for the children to improve their physical fitness. Question: Will children with heart disease have improved their physical condition three months after a stay at Geilomo?

Work schedule: The project will have a duration of 3 years. The project will seek approval of the Regional Committee for Medical Research Ethics in May 2012. Interview Guide, information sheet and consent form has been prepared. Data collection for the study 2AB can start in March 2013. The first interviews will be conducted after 3 months, in June 2013. Data collection is expected to be completed in December 2013. The analysis will take place in parallel with the interview work. In 2014 and 2015 completed the writing of articles (3 pieces) and publication of results.

Method: In order to shed light on the problem in study 1, the investigators will use semi-structured interview. 16 children and 16 parents to be interviewed after 3 months. Study 2a) To get information about their child's activity level in the home environment the investigators will use structured questionnaires. It is one form for children (36 persons) and another form for their parents (36 persons). Study 2b) All children (36 persons) conducting physical fitness test at the first visit and after three months. Children can be referred from across the country via the referral form. Dr. Henrik Holm (OUS) and Dr. Asle Hirth (HUS) determines participation according to inclusion and exclusion criteria.

Parents submit a written consent on behalf of themselves and their children.

Scientific significance: This application describes two related studies, both of which are expected to provide important information that can provide better services for children with heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Children with heart disease in the age groups 6-7 years and 11-12 years with the need for lifelong medical treatment.

Exclusion Criteria:

* Children with serious mentally retardation and/or significant physical disabilities. Children and caregivers who does not speak norwegian or for other reasons have problems with communication that makes a interview difficult.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Increased level of physical activity | 3 months

SECONDARY OUTCOMES:
Increased physical fitness | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Geilomo barnesykehus, Geilo, Buskerud, Norway